CLINICAL TRIAL: NCT05078346
Title: Observational Study to Determine the Association Between Self-rated, Perceived Immune Fitness (Using Questionnaire) With Biological Assessment of Immune Fitness (Immune Signatures in the Blood).
Brief Title: Immune Fitness Prediction
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024_NR
Record Dates: First submitted 2021-08-26; First posted 2021-10-14 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Healthy Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall objective of the study is to determine whether self-rated, perceived immune fitness (using questionnaire) is associated with biological assessment of immune fitness (immune signatures in the blood).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and sign the informed consent
2. Healthy adult men and/or women, 35-65 years old
3. BMI >18 and <30 kg/m2

Exclusion Criteria:

1. Volunteer who cannot be expected to comply with the protocol
2. Individuals with self-reported chronic disease; or who have any clinical condition which the investigator deems relevant for exclusion from the study,
3. Individuals with an impaired immune system that may confound immune response testing; i.e. any condition that impairs participant immune response through either the condition itself or through the treatment of the condition,
4. Family or hierarchical relationships with Clinical Innovation Lab at Nestlé Research, Lausanne, Switzerland

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Percentage of different immune cell types in whole blood | 6 - 12 months after the start of the trial
  Immune cell type profiling in whole blood by mass cytometry
Relative quantification of immune protein in plasma | 6 - 12 months after the start of the trial
  Proteomic analysis in plasma by proximity extension assay
Amount of cytokines expressed by peripheral blood mononuclear cells | 6 - 12 months after the start of the trial
  Cytokine quantification by proximity extension assay
Amount of analytes in serum | 6 - 12 months after the start of the trial
  Blood chemistry

CONTACTS AND LOCATIONS:
Locations (1):
- Nestlé Clinical Research Unit, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided